CLINICAL TRIAL: NCT06970704
Title: Erector Spinae Plane Block Combined With General Anesthesia Versus General Anesthesia Alone in Spine Surgeries for Postoperative Pain, A Randomized Controlled Trial
Brief Title: Erector Spinae Plane Block in Spine Surgeries for Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMASU MS 681/2023
Record Dates: First submitted 2024-10-01; First posted 2025-05-14 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-09

CONDITIONS: Spine Fusion; Spine Metastases; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Erector Spinae Plane Block (ESPB) (Study) (Active Comparator): Patients in this group will receive Erector Spinae Plane Block (20 ml bupivacaine 0.25%) combined with general anesthesia
  Interventions: Other: Erector Spinae Plane Block using 0.25 % bupivacaine
- Group General Anesthesia (GA) (Control) (Active Comparator): Patients in this group will receive conventional general anesthesia
  Interventions: Other: Erector Spinae Plane Block using 0.25 % bupivacaine

INTERVENTIONS:
Other: Erector Spinae Plane Block using 0.25 % bupivacaine — After induction of anesthesia and prone positioning and before surgery, Erector Spinae Plane Block was performed bilaterally using a low-frequency curved ultrasound transducer placed in a longitudinal orientation 3 cm lateral to the spinous process one vertebral level above a predetermined marked surgical incision. An 8-cm 22-gauge block needle was inserted in a cephalad to caudad direction until the tip lay in the interfascial plane below the erector spinae muscle, the block was performed by injection of 20 ml of 0.25% bupivacaine. Fentanyl 1 µg/kg as a rescue analgesia was given based on hemodynamic parameters.

SUMMARY:
This prospective single-blind randomized controlled study on 50 patients between 18 and 65 years, both sexes, with ASA I-II and undergoing elective lumbar spine surgical procedures. They were equally divided into two groups: Group Erector Spinae Plane Block (ESPB) (Study): (number = 25) received Erector Spinae Plane Block (20 ml bupivacaine 0.25%) combined with general anesthesia. Group General Anesthesia (GA) (Control): (number = 25) received conventional general anesthesia.

DETAILED DESCRIPTION:
In both groups, on arrival to the operation room, a multi-channel monitor will be attached to the patient to display continuous electrocardiogram (ECG) monitoring, heart rate (HR), non-invasive blood pressure, pulse oximeter, temperature probe, capnogram, and anesthetic gas analysis. An intravenous line will be secured, then lactated Ringer's solution will be started at 5 ml/kg/h. Ten minutes before induction of anesthesia, all patients will be premedicated with intravenous midazolam 0.02 mg/kg. Patients will be preoxygenated with 100% oxygen for 3 minutes. In both groups, induction of anesthesia will be carried out by intravenous administration of fentanyl 1 µg/kg, lidocaine 1.5 mg/kg, and propofol 2 mg/kg. After loss of verbal communication, 0.5 mg/kg atracurium will be administered. Intermittent positive pressure ventilation will be adjusted to maintain an end-tidal carbon dioxide partial pressure between 30 and 35 mmHg. Anesthesia will be maintained with 1-2% isoflurane, 0.1 mg/kg atracurium bolus doses will be administered every 20 minutes, and 0.5 µg/kg fentanyl will be administered every 30 minutes.

In the Erector Spinae Plane block (ESPB) group, after prone positioning and before surgery, Erector Spinae Plane Block will be performed bilaterally using a low-frequency curved ultrasound transducer placed in a longitudinal orientation 3 cm lateral to the spinous process one vertebral level above a predetermined marked surgical incision. An 8-cm 22-gauge block needle will be inserted in a cephalad to caudad direction until the tip lies in the interfascial plane below the erector spinae muscle; the block will be performed by injection of 20 ml of 0.25% bupivacaine. In both groups, fentanyl 1 µg/kg as rescue analgesia will be given based on hemodynamic parameters.

If the mean arterial blood pressure (MAP) has fallen below 65 mmHg, 5 mg of ephedrine will be administered, and an intravenous bolus of 0.5 mg of atropine will be administered in case of bradycardia if the heart rate ≤50 bpm. The blood pressure will return to the baseline value before surgical field closure. Then at the end of surgery, the isoflurane vaporizer will be turned off, and the muscle relaxant will be reversed with neostigmine 0.04 mg/kg and atropine 0.02 mg/kg. The endotracheal tube will be removed after the patient regains consciousness and full muscle power, breathes spontaneously, and responds to verbal commands. Isoflurane consumption was measured at the end of surgery.

Postoperative pain management:

A standardized analgesic regimen will be prescribed in the postoperative period. All patients will receive 1 gm of paracetamol every 6 h. If the numeric rating scale (NRS) is more than 3, intravenous morphine 3mg will be administered by an investigator blinded to group assignment.

Clinical evaluation:

Total intravenous drug administration at the post-anesthesia care unit (PACU) and over the 48 hours was recorded. Opioid-related adverse events arising from the analgesic protocol will be systematically assessed at the PACU and surgical ward. The presence of nausea, vomiting, respiratory depression, pruritus, urinary retention requiring evacuation, allergy, and hallucinations will be recorded as binary (yes/no). Arterial oxygen saturation (pulse oximetry), heart and respiratory rates, and blood pressure will also be recorded every 6 hours.

The Ramsay Sedation Scale will be assessed postoperatively. The Ramsay sedation scale comprises two clearly defined groups of scores: those of 1, 2, and 3 are given in assessing degrees of wakefulness, and those of 4, 5, and 6 are given in assessing degrees of sleep. The six levels of the Ramsay sedation scale allow for visual assessments of sedation in patients who are responsive to such assessments

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged from 18 and 65 years, both sexes
2. The American Society of Anesthesiology (ASA) physical status I-II
3. Scheduled for elective lumbar spine surgical procedures

Exclusion Criteria:

1. Coagulation disorders
2. BMI > 30 or < 18 kg/m2
3. Patients with surgical site infection
4. Known sensitivity or contraindication to local anesthetics
5. History of psychological disorders
6. Patients with unstable spine integrity like fractures or scoliosis
7. Hypertensive, cardiac, and diabetic patients,
8. Known alcohol or substance abuse within the last 6 months and Daily opioid intake

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-12-31 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Postoperative pain severity | Postoperatively Day 1
  Using Pain Numeric Rating Scale Scores
Time to the first postoperative rescue analgesic | Postoperatively Day 1
  Time to first use of morphine
Fentanyl consumption. | During Intraoperative period
  Intraoperative fentanyl consumption
Isoflurane consumption. | During Intraoperative period
  Intraoperative fentanyl and isoflurane consumption.

SECONDARY OUTCOMES:
Changes in mean arterial pressure | Immediately before the operation till Postoperatively Day 1
  Perioperative changes in mean arterial pressure
Changes in heart rate | Immediately before the operation till Postoperatively Day 1
  Perioperative changes in heart rate
Postoperative nausea and vomiting | Postoperatively Day 1
  Number of postoperative nausea and vomiting episodes

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Prabhakar NK, Chadwick AL, Nwaneshiudu C, Aggarwal A, Salmasi V, Lii TR, Hah JM. Management of Postoperative Pain in Patients Following Spine Surgery: A Narrative Review. Int J Gen Med. 2022 May 2;15:4535-4549. doi: 10.2147/IJGM.S292698. eCollection 2022. PMID 35528286
- [Background] Ye Y, Bi Y, Ma J, Liu B. Thoracolumbar interfascial plane block for postoperative analgesia in spine surgery: A systematic review and meta-analysis. PLoS One. 2021 May 21;16(5):e0251980. doi: 10.1371/journal.pone.0251980. eCollection 2021. PMID 34019598
- [Background] Hyland SJ, Brockhaus KK, Vincent WR, Spence NZ, Lucki MM, Howkins MJ, Cleary RK. Perioperative Pain Management and Opioid Stewardship: A Practical Guide. Healthcare (Basel). 2021 Mar 16;9(3):333. doi: 10.3390/healthcare9030333. PMID 33809571
- [Background] Jin Y, Zhao S, Cai J, Blessing M, Zhao X, Tan H, Li J. Erector Spinae Plane Block for Perioperative Pain Control and Short-term Outcomes in Lumbar Laminoplasty: A Randomized Clinical Trial. J Pain Res. 2021 Sep 3;14:2717-2727. doi: 10.2147/JPR.S321514. eCollection 2021. PMID 34512011
- [Background] Rasheed AM, Amirah MF, Abdallah M, P J P, Issa M, Alharthy A. Ramsay Sedation Scale and Richmond Agitation Sedation Scale: A Cross-sectional Study. Dimens Crit Care Nurs. 2019 Mar/Apr;38(2):90-95. doi: 10.1097/DCC.0000000000000346. PMID 30702478
- [Background] Nashibi M, Sezari P, Safari F, Teymourian H, Asgari S, Mottaghi K. The effect of erector spinae plane block on the use of anesthetic medications in lumbar spine surgery. Agri. 2023 Oct;35(4):228-235. doi: 10.14744/agri.2022.48992. PMID 37886866
- [Background] Elewa AM, Faisal M, Sjoberg F, Abuelnaga ME. Comparison between erector spinae plane block and paravertebral block regarding postoperative analgesic consumption following breast surgery: a randomized controlled study. BMC Anesthesiol. 2022 Jun 18;22(1):189. doi: 10.1186/s12871-022-01724-3. PMID 35717148
- [Background] Zhang Q, Wu Y, Ren F, Zhang X, Feng Y. Bilateral ultrasound-guided erector spinae plane block in patients undergoing lumbar spinal fusion: A randomized controlled trial. J Clin Anesth. 2021 Feb;68:110090. doi: 10.1016/j.jclinane.2020.110090. Epub 2020 Oct 20. PMID 33096517